CLINICAL TRIAL: NCT02396212
Title: An Open-label, Single-arm, Active-treatment, Efficacy and Safety Study of Canakinumab (ACZ885) Administered for at Least 48 Weeks in Japanese Patients With Systemic Juvenile Idiopathic Arthritis (SJIA)
Brief Title: Study of Efficacy and Safety of Canakinumab in Japanese Patients With SJIA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885G1301; 2018-002355-15 (EudraCT Number)
Record Dates: First submitted 2015-02-25; First posted 2015-03-24 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Systemic Juvenile Idiopathic Arthritis
Keywords: ACZ885; canakinumab; Juvenile Rheumatoid arthritis (JRA) chronic; systemic inflammatory disorder; painful joints; inflammation of the synovial membrane; auto-immune rheumatoid disease; reactive rheumatoid arthritis; Systemic Juvenile Rheumatoid arthritis (SJRA); Japanese patients
MeSH Terms: conditions — Arthritis, Juvenile; Bronchiolitis Obliterans Syndrome; Arthralgia; Rheumatoid Arthritis, Systemic Juvenile | interventions — canakinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Canakinumab (Experimental): All patients received canakinumab (ACZ885) as open-label study medication. Patients were administered canakinumab 4 mg/kg every 4 weeks. The maximal total single dose of canakinumab allowed was 300 mg.
  Interventions: Biological: Canakinumab

INTERVENTIONS:
Biological: Canakinumab — canakinumab was provided as a 150 mg/1 mL solution for subcutaneous injection and administered at 4mg/kg every 4 weeks.
  Other Names: ACZ885

SUMMARY:
This was a phase III study designed to provide efficacy and safety data for canakinumab administered for at least 48 weeks as subcutaneous (s.c.) injection every 4 weeks (q4wk) in Japanese patients with Systemic Juvenile Idiopathic Arthritis (SJIA). Interim analysis (IA) data at Week 28 and 48 from this study supported a registration submission of canakinumab in the indication of SJIA in Japan.

ELIGIBILITY:
Inclusion Criteria

- Confirmed diagnosis of SJIA as per International League Against Rheumatism (ILAR) definition (Petty, et al. 2004) that must have occurred at least 3 months prior to enrollment with an onset of disease < 16 years of age: Arthritis in one or more joints, with or preceded by fever of at least 2 weeks duration that is documented to be daily/quotidian for at least 3 days and accompanied by one or more of the following: Rash due to SJIA, lymphadenopathy, Hepatomegaly/Splenomegaly, Serositis

* Active disease at the time of baseline defined as follows:
* At least 2 joints with active arthritis
* Documented spiking, intermittent fever (body temperature > 38°C) for at least 1 day during the screening epoch and within 1 week before first canakinumab dose
* C-Reactive Protein (CRP) > 30 mg/L(3 mg/dL) (normal range < 10 mg/L(1 mg/dL))
* Negative TB screen (Chest X-ray and T-SPOT test)

Exclusion Criteria:

* With active or recurrent bacterial, fungal or viral infection at the time of enrollment, including patients with evidence of Human Immunodeficiency Virus (HIV) infection, Hepatitis B and Hepatitis C infection. Patients with resolved/previous hepatitis B infection (a negative HBs antigen, but a positive anti-HBs antibody and/or anti-HBc antibody).
* With underlying metabolic, renal, hepatic, infectious or gastrointestinal conditions which in the opinion of the investigator immunocompromises the patient and /or places the patient at unacceptable risk for participation.
* With neutropenia (absolute neutrophil count < 1500/mm3) at screening.

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Japan (6):
  - Novartis Investigative Site, Ōbu, Aichi-ken
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: http://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Nishimura K, Hara R, Umebayashi H, Takei S, Iwata N, Imagawa T, Shimizu M, Tomiita M, Seko N, Kitawaki T, Yokota S. Efficacy and safety of canakinumab in systemic juvenile idiopathic arthritis: 48-week results from an open-label phase III study in Japanese patients. Mod Rheumatol. 2021 Jan;31(1):226-234. doi: 10.1080/14397595.2020.1783163. Epub 2020 Jul 29. PMID 32552266

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned to enroll approximately 20 patients in this study. There were19 patients enrolled and data from all patients were analyzed.
Groups:
- Canakinumab 4 mg/kg Every 4 Weeks: All patients received canakinumab (ACZ885) as open-label study medication. Patients were administered canakinumab 4 mg/kg every 4 weeks. The maximal total single dose of canakinumab allowed was 300 mg.
Period: Overall Study
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Started | 19
Completed | 16
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.9 (4.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Minimum Adapted American College of Rheumatology (ACR) Pediatric 30 Criteria
Description: Minimum Adapted ACR Pediatric 30 criteria is defined as improvement from baseline at least 30% in at least 3 of response variables 1 to 6 in Adapted ACR Pediatric response variables and no intermittent fever (i.e. axillary, oral, or rectal body temperature ≤ 38°C) in the preceding week (variable 7), with no more than one variable 1-6 worsening by more than 30%. Adapted ACR Pediatric response variables consists of following 7 variables: 1. Physician's Global Assessment of disease activity on a 0-100 mm VAS; 2. Parent's or Patient's (if appropriate in age) Global Assessment of Patient's overall wellbeing based upon the 0-100 mm VAS in the Child Health Assessment Questionnaire (CHAQ); 3. Functional ability: CHAQ; 4. Number of joints with active arthritis; 5. Number of joints with limitation of motion; 6. Laboratory measure of inflammation: CRP (mg/L); 7. Absence of intermittent fever due to SJIA during the preceding week.
Time Frame: Week 8
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
Percentage of Participants | 100.0

2. Primary Outcome: Percentage of Participants With Canakinumab Treatment Who Were Able to Taper Corticosteroids Successfully
Description: To evaluate the percentage of participants with canakinumab treatment who were able to taper corticosteroids successfully at Week 28
Time Frame: Week 28
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Number; unit: Percentage of Participants
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
Percentage of Participants | 73.7

3. Secondary Outcome: Percentage of Participants Who Met the Adapted ACR Pediatric 30/50/70/90/100 Criteria of Canakinumab Over Time
Description: Adapted ACR Pediatric 30/50/70/90/100 criteria was assessed based on the following 7 variables: 1. Physician's Global Assessment of disease activity on a 0-100 mm VAS; 2. Parent's or Patient's (if appropriate in age) Global Assessment of Patient's overall wellbeing based upon the 0-100 mm VAS in the CHAQ; 3. Functional ability: CHAQ; 4. Number of joints with active arthritis; 5. Number of joints with limitation of motion; 6. Laboratory measure of inflammation: CRP (mg/L); 7. Absence of intermittent fever due to SJIA during the preceding week. Response was defined as more than or equal to (≥) 30%/50%/70%/90% or 100% improvement in at least 3 of 6 response variables and no intermittent fever in the preceding week (variable 7) with no more than one variable 1-6 worsening by more than 30%.
Time Frame: Weeks 4, 8, 28, 48, 96, 144, end of study (EOS) (up to Week 164)
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Number; unit: Percentage of Participants
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
Percentage of Participants
  Week 4 adapted ACR Pediatric 30 | 94.7
  Week 4 adapted ACR Pediatric 50 | 94.7
  Week 4 adapted ACR Pediatric 70 | 94.7
  Week 4 adapted ACR Pediatric 90 | 84.2
  Week 4 adapted ACR Pediatric 100 | 47.4
  Week 8 adapted ACR Pediatric 30 | 100.0
  Week 8 adapted ACR Pediatric 50 | 100.0
  Week 8 adapted ACR Pediatric 70 | 100.0
  Week 8 adapted ACR Pediatric 90 | 89.5
  Week 8 adapted ACR Pediatric 100 | 68.4
  Week 28 adapted ACR Pediatric 30: number analyzed (Participants) | 16
  Week 28 adapted ACR Pediatric 30 | 100.0
  Week 28 adapted ACR Pediatric 50: number analyzed (Participants) | 16
  Week 28 adapted ACR Pediatric 50 | 100.0
  Week 28 adapted ACR Pediatric 70: number analyzed (Participants) | 16
  Week 28 adapted ACR Pediatric 70 | 100.0
  Week 28 adapted ACR Pediatric 90: number analyzed (Participants) | 16
  Week 28 adapted ACR Pediatric 90 | 100.0
  Week 28 adapted ACR Pediatric 100: number analyzed (Participants) | 16
  Week 28 adapted ACR Pediatric 100 | 56.3
  Week 48 adapted ACR Pediatric 30: number analyzed (Participants) | 16
  Week 48 adapted ACR Pediatric 30 | 100.0
  Week 48 adapted ACR Pediatric 50: number analyzed (Participants) | 16
  Week 48 adapted ACR Pediatric 50 | 100.0
  Week 48 adapted ACR Pediatric 70: number analyzed (Participants) | 16
  Week 48 adapted ACR Pediatric 70 | 100.0
  Week 48 adapted ACR Pediatric 90: number analyzed (Participants) | 16
  Week 48 adapted ACR Pediatric 90 | 87.5
  Week 48 adapted ACR Pediatric 100: number analyzed (Participants) | 16
  Week 48 adapted ACR Pediatric 100 | 68.8
  Week 96 adapted ACR Pediatric 30: number analyzed (Participants) | 16
  Week 96 adapted ACR Pediatric 30 | 100.0
  Week 96 adapted ACR Pediatric 50: number analyzed (Participants) | 16
  Week 96 adapted ACR Pediatric 50 | 100.0
  Week 96 adapted ACR Pediatric 70: number analyzed (Participants) | 16
  Week 96 adapted ACR Pediatric 70 | 100.0
  Week 96 adapted ACR Pediatric 90: number analyzed (Participants) | 16
  Week 96 adapted ACR Pediatric 90 | 93.8
  Week 96 adapted ACR Pediatric 100: number analyzed (Participants) | 16
  Week 96 adapted ACR Pediatric 100 | 62.5
  Week 144 adapted ACR Pediatric 30: number analyzed (Participants) | 5
  Week 144 adapted ACR Pediatric 30 | 100.0
  Week 144 adapted ACR Pediatric 50: number analyzed (Participants) | 5
  Week 144 adapted ACR Pediatric 50 | 100.0
  Week144 adapted ACR Pediatric 70: number analyzed (Participants) | 5
  Week144 adapted ACR Pediatric 70 | 100.0
  Week 144 adapted ACR Pediatric 90: number analyzed (Participants) | 5
  Week 144 adapted ACR Pediatric 90 | 100.0
  Week 144 adapted ACR Pediatric 100: number analyzed (Participants) | 5
  Week 144 adapted ACR Pediatric 100 | 80.0
  Week EOS adapted ACR Pediatric 30 | 89.5
  End of Study (EOS) adapted ACR Pediatric 50 | 89.5
  EOS adapted ACR Pediatric 70 | 89.5
  EOS adapted ACR Pediatric 90 | 84.2
  EOS adapted ACR Pediatric 100 | 63.2

4. Secondary Outcome: Absolute Change From Baseline in the Adapted ACR Pediatric Criteria of Canakinumab Over Time: ACR Component: Physician's Global Assessment of Disease Activity
Description: ACR component, Physician's Global Assessment of disease activity on a 0 - 100 mm VAS by visit is the first response ACR variable in the ACR pediatric criteria. The VAS scale ranges from no disease activity (0 mm) to very severe disease activity (100 mm). Lower scale indicates decreased disease activity. Change from baseline was calculated by subtracting baseline value from post baseline value.
Time Frame: Baseline, Weeks 4, 8, 28, 48, 96, 144, EOS (up to Week 164)
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
units on a scale
  Week 4 | -60.2 (32.27)
  Week 8 | -62.2 (28.23)
  Week 28: number analyzed (Participants) | 16
  Week 28 | -62.2 (28.61)
  Week 48: number analyzed (Participants) | 16
  Week 48 | -63.9 (28.81)
  Week 96: number analyzed (Participants) | 16
  Week 96 | -63.1 (26.99)
  Week 144: number analyzed (Participants) | 5
  Week 144 | -61.0 (37.24)
  EOS | -61.4 (31.05)

5. Secondary Outcome: Absolute Change From Baseline in the Adapted ACR Pediatric Criteria of Canakinumab Over Time: ACR Component: CHAQ: Parent's or Patient's Global Assessment of Patient's Overall Well-being as Part of CHAQ
Description: ACR component, Parent's or Patient's (if appropriate in age)Global Assessment of patient's overall well-being as part of CHAQ on a 0 - 100 mm VAS by visit is the second response variable in the ACR pediatric criteria. The VAS scale ranges from 0-100 mm, from very well (0 mm) to very poor (100 mm). Lower scale indicates improvement of patient's overall well-being. Absolute change is calculated by subtracting baseline value from post baseline value.
Time Frame: Baseline, Weeks 4, 8, 28, 48, 96, 144, EOS up to Week 164
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
units on a scale
  Week 4 | -64.4 (40.80)
  Week 8 | -73.5 (24.05)
  Week 28: number analyzed (Participants) | 16
  Week 28 | -71.9 (23.13)
  Week 48: number analyzed (Participants) | 16
  Week 48 | -68.6 (28.67)
  Week 96: number analyzed (Participants) | 16
  Week 96 | -68.4 (27.72)
  Week 144: number analyzed (Participants) | 5
  Week 144 | -72.8 (25.65)
  EOS | -68.1 (26.29)

6. Secondary Outcome: Absolute Change From Baseline in the Adapted ACR Pediatric Criteria of Canakinumab Over Time: ACR Component: CHAQ: Functional Ability Score
Description: Disability Score as part of CHAQ per functional ability score (range from 0 to 3) is one of the variable in the ACR ped criteria. The CHAQ was used to assess physical ability & functional status of patients as well as quality of life. The disability dimension consists of 20 multiple choice items concerning difficulty in performing 8 common activity categories of daily living: dressing & grooming, arising, eating, walking, reaching, personal hygiene, gripping & other "activities". Subjects choose from 4 responses, ranging from 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty) & 3 (unable to do). Standard Disability Index (SDI) was computed by summing up the computed scores for each activity category and dividing by the number of categories answered. The lower the response the more positive the results & the higher the response, the less positive the results. Change from baseline was calculated by subtracting baseline value from post baseline value.
Time Frame: Baseline, Weeks 4, 8, 28, 48, 96, 144, EOS (up to Week 164)
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
units on a scale
  Week 4 | -0.833 (0.7750)
  Week 8 | -0.912 (0.7338)
  Week 28: number analyzed (Participants) | 16
  Week 28 | -0.998 (0.7871)
  Week 48: number analyzed (Participants) | 16
  Week 48 | -1.013 (0.7963)
  Week 96: number analyzed (Participants) | 16
  Week 96 | -0.951 (0.8381)
  Week 144: number analyzed (Participants) | 5
  Week 144 | -1.026 (0.9465)
  EOS | -0.938 (0.7682)

7. Secondary Outcome: Absolute Change From Baseline in the Adapted ACR Pediatric Criteria of Canakinumab Over Time: ACR Component: Number of Joints With Active Arthritis
Description: ACR component, Number of joints with active arthritis was assessed as the forth response variables of ACR Pediatric Criteria.
Time Frame: Baseline, Weeks 4, 8, 28, 48, 96, 144, EOS (up to Week 164)
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
joints
  Week 4 | -5.2 (4.87)
  Week 8 | -6.2 (7.71)
  Week 28: number analyzed (Participants) | 16
  Week 28 | -4.4 (3.44)
  Week 48: number analyzed (Participants) | 16
  Week 48 | -4.4 (3.44)
  Week 96: number analyzed (Participants) | 16
  Week 96 | -4.4 (3.18)
  Week 144: number analyzed (Participants) | 5
  Week 144 | -5.2 (2.68)
  EOS | -5.6 (8.10)

8. Secondary Outcome: Absolute Change From Baseline in the Adapted ACR Pediatric Criteria of Canakinumab Over Time: ACR Component: Number of Joints With Limitation of Motion
Description: ACR component, Number of joints with limitation of motion is the fifth response variable in the ACR ped criteria.
Time Frame: Baseline, Weeks 4, 8, 28, 48, 96, 144, EOS (up to Week 164)
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
joints
  Week 4 | -3.9 (4.02)
  Week 8 | -4.2 (4.30)
  Week 28: number analyzed (Participants) | 16
  Week 28 | -3.4 (3.79)
  Week 48: number analyzed (Participants) | 16
  Week 48 | -3.5 (3.78)
  Week 96: number analyzed (Participants) | 16
  Week 96 | -3.4 (3.59)
  Week 144: number analyzed (Participants) | 5
  Week 144 | -3.8 (2.86)
  EOS | -3.7 (4.81)

9. Secondary Outcome: Number of Participants Having Fever in the Adapted ACR Pediatric Criteria of Canakinumab Over Time
Description: ACR component, Number of participants having fever is the seventh response variable in the ACR ped criteria.
Time Frame: Baseline, Day 3, Weeks 2, 8, 28, 48, 56, 96, 124, 144, EOS (up to Week 164)
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Number; unit: participants
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
participants
  Baseline | 19
  Day 3 | 16
  Week 2 | 2
  Week 8 | 0
  Week 28: number analyzed (Participants) | 16
  Week 28 | 0
  Week 48: number analyzed (Participants) | 16
  Week 48 | 0
  Week 56: number analyzed (Participants) | 16
  Week 56 | 1
  Week 96: number analyzed (Participants) | 16
  Week 96 | 0
  Week 124: number analyzed (Participants) | 8
  Week 124 | 1
  Week 144: number analyzed (Participants) | 5
  Week 144 | 0
  EOS | 0

10. Secondary Outcome: Percentage Change From Baseline in the Adapted ACR Pediatric Criteria of Canakinumab Over Time: ACR Component: Standardized C-Reactive Protein (CRP)
Description: ACR component, Standardized CRP is the sixth response variable in the ACR ped criteria. CRP values were standardized to a normal range of 0 to 10 mg/L.
Time Frame: Baseline, Weeks 4, 8, 28, 48, 96, 144, EOS (up to Week 164)
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
Percentage change
  Week 4 | -89.45 (41.431)
  Week 8 | -96.95 (6.915)
  Week 28: number analyzed (Participants) | 16
  Week 28 | -98.19 (2.567)
  Week 48: number analyzed (Participants) | 16
  Week 48 | -97.64 (6.333)
  Week 96: number analyzed (Participants) | 16
  Week 96 | -97.95 (3.730)
  Week 144: number analyzed (Participants) | 5
  Week 144 | -98.58 (1.330)
  EOS | -89.71 (20.717)

11. Secondary Outcome: Percentage of Participants Who Had Flares With Canakinumab Treatment Over Time
Description: Flare was defined by at least 1 of the following: Reappearance of SJIA-related (e.g., not due to infection) fever (> 38°C) lasting for at least 2 consecutive days &/OR Flare according to the JIA pediatric criteria for flare (all criteria must be met): ≥ 30% worsening in at least 3 of the 6 response variables and ≥ 30% improvement in at not more than 1 of the 6 response variables if the physician's or parent's global assessment is 1of 3 response variables used to define flare, worsening of ≥ 20 mm must be present, if the number of active joints or joints with limitation of motion is one of 3 response variables used to define flare, worsening in ≥ 2 joints must be present if CRP is used to define flare, CRP must be > 30 mg/L
Time Frame: > Day3, to <= Week 124
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
Percentage of participants
  >Day 3 =<Week 2 | 5.3
  >Week 2 =<Week 4 | 5.3
  >Week 4 =<Week 8 | 5.3
  >Week 8 =<Week 12: number analyzed (Participants) | 18
  >Week 8 =<Week 12 | 5.6
  >Week 12 =<Week 16: number analyzed (Participants) | 18
  >Week 12 =<Week 16 | 5.6
  >Week 92 =<Week 96: number analyzed (Participants) | 16
  >Week 92 =<Week 96 | 6.3
  >Week 104 =<Week 108: number analyzed (Participants) | 13
  >Week 104 =<Week 108 | 7.7
  >Week 120 =<Week 124: number analyzed (Participants) | 8
  >Week 120 =<Week 124 | 12.5

12. Secondary Outcome: Percentage of Participants Who Achieved Inactive Disease (With and Without Duration of Morning Stiffness) With Canakinumab Treatment Over Time
Description: Inactive disease was defined as meeting all of the following: No joints with active arthritis; No fever (body temperature ≤ 38°C); No rheumatoid rash, serositis, splenomegaly, hepatomegaly or generalized lymphadenopathy attributable to JIA; Normal CRP; Physician's global assessment of disease activity score ≤ 10 mm
Time Frame: Weeks 4, 8, 28, 48, 96, 144, EOS (up to Week 164)
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Number; unit: Percentage of participants
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
Percentage of participants
  Week 4 | 63.2
  Week 8 | 63.2
  Week 28: number analyzed (Participants) | 16
  Week 28 | 75.0
  Week 48: number analyzed (Participants) | 16
  Week 48 | 75.0
  Week 96: number analyzed (Participants) | 16
  Week 96 | 75.0
  Week 144: number analyzed (Participants) | 5
  Week 144 | 80.0
  EOS | 68.4

13. Secondary Outcome: Percentage of Participants With Canakinumab Treatment Who Were Able to Taper Corticosteroids Successfully Over Time
Description: To evaluate the percentage of participants with canakinumab treatment who were able to taper corticosteroids successfully over time
Time Frame: Weeks 28, 48, 96, 144, EOS (up to Week 164)
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Number; unit: percentage of perticipants
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
percentage of perticipants
  Week 28: number analyzed (Participants) | 16
  Week 28 | 87.5
  Week 48: number analyzed (Participants) | 16
  Week 48 | 81.3
  Week 96: number analyzed (Participants) | 16
  Week 96 | 87.5
  Week 144: number analyzed (Participants) | 5
  Week 144 | 100.0
  EOS: number analyzed (Participants) | 18
  EOS | 66.7

14. Secondary Outcome: Absolute Change From Baseline of Corticosteroids Dose Reduction With Canakinumab Treatment Over Time
Description: To evaluate the change from baseline of corticosteroids dose reduction with canakinumab treatment over time
Time Frame: Baseline, Weeks 28, 48, 96, 144, EOS (up to Week 164)
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
mg/kg/day
  Week 28: number analyzed (Participants) | 16
  Week 28 | -0.133 (0.1676)
  Week 48: number analyzed (Participants) | 16
  Week 48 | -0.195 (0.2317)
  Week 96: number analyzed (Participants) | 16
  Week 96 | -0.226 (0.2618)
  Week 144: number analyzed (Participants) | 5
  Week 144 | -0.296 (0.2545)
  EOS: number analyzed (Participants) | 18
  EOS | -0.171 (0.2334)

15. Secondary Outcome: Serum Concentration of Canakinumab
Description: To evaluate serum concentration (mean, standard deviation) of canakinumab.
Time Frame: Baseline, Weeks 4, 24, 48, 72, 96, EOS (up to Week 164)
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
μg/mL
  Baseline | 0.01 (0.05)
  Week 4 | 15.7 (5.19)
  Week 24: number analyzed (Participants) | 16
  Week 24 | 31.3 (11.5)
  Week 48: number analyzed (Participants) | 16
  Week 48 | 31.1 (9.08)
  Week 72: number analyzed (Participants) | 16
  Week 72 | 30.6 (8.95)
  Week 96: number analyzed (Participants) | 16
  Week 96 | 29.5 (8.49)
  EOS | 28.3 (6.41)

16. Secondary Outcome: Pharmacodynamics (PD) Assessment: Total IL-1 Beta
Description: To evaluate serum total IL-1 Beta concentration by visit.
Time Frame: Baseline, Weeks 4, 24, 48, 72, 96, EOS (up to Week 164)
Population: The FAS consisted of all 19 patients who were enrolled and received at least one dose of canakinumab.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
Number analyzed (Participants) | 19
pg/mL
  Baseline | 0.72 (0.97)
  Week 4 | 49.8 (36.3)
  Week 24: number analyzed (Participants) | 16
  Week 24 | 85.2 (61.6)
  Week 48: number analyzed (Participants) | 16
  Week 48 | 81.2 (62.0)
  Week 72: number analyzed (Participants) | 16
  Week 72 | 75.3 (36.6)
  Week 96: number analyzed (Participants) | 16
  Week 96 | 74.4 (35.9)
  EOS | 101 (89.1)

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV) up to approximately 39 months.
Arm/Group | Canakinumab 4 mg/kg Every 4 Weeks
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 10/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab 4 mg/kg Every 4 Weeks (N=19)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 3
Adrenal insufficiency (Endocrine disorders) | 2
Pyrexia (General disorders) | 2
Epstein-Barr virus infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Varicella (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Still's disease (Musculoskeletal and connective tissue disorders) | 6
Altered state of consciousness (Nervous system disorders) | 1
Somatic symptom disorder (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canakinumab 4 mg/kg Every 4 Weeks (N=19)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Motion sickness (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Chalazion (Eye disorders) | 1
Conjunctivitis allergic (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 6
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Injection site pain (General disorders) | 1
Injection site reaction (General disorders) | 5
Malaise (General disorders) | 1
Pyrexia (General disorders) | 1
Vessel puncture site pain (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 5
Hepatic steatosis (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Allergy to arthropod sting (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Angular cheilitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 6
Gastroenteritis viral (Infections and infestations) | 2
Herpes zoster (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 4
Impetigo (Infections and infestations) | 1
Influenza (Infections and infestations) | 4
Lice infestation (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 12
Otitis media acute (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 4
Viral infection (Infections and infestations) | 1
Viral pharyngitis (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 2
Arthropod sting (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 4
Alanine aminotransferase increased (Investigations) | 4
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood creatine phosphokinase decreased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Intraocular pressure increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Hyperalbuminaemia (Metabolism and nutrition disorders) | 2
Hyperamylasaemia (Metabolism and nutrition disorders) | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Still's disease (Musculoskeletal and connective tissue disorders) | 2
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Histiocytic necrotising lymphadenitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 6
Neuropathy peripheral (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Blister (Skin and subcutaneous tissue disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Eczema (Skin and subcutaneous tissue disorders) | 4
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Macule (Skin and subcutaneous tissue disorders) | 1
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2014-11-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT02396212/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT02396212/SAP_001.pdf